CLINICAL TRIAL: NCT04605484
Title: Phase 2 Multicenter, Randomized, Double-blind, Placebo-controlled, Multiple Dosing Interval, 2-period Study of the Safety, Tolerability and Effectiveness of Adoptively Transferred Posoleuccel (ALVR105) Multivirus-specific T Cells in Kidney Transplant Recipients With Either High or Low Levels of BK Viremia
Brief Title: Study of Posoleucel (Formerly Known as ALVR105; Viralym-M) in Kidney Transplant Patients With BK Viremia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlloVir (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P-105-201
Record Dates: First submitted 2020-10-15; First posted 2020-10-28 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: BK Virus Nephropathy; BK Virus Infection
MeSH Terms: interventions — Cell Count

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Posoleucel (Experimental): Arm 1: Regimen A
  Interventions: Biological: Posoleucel (formerly known as ALVR105) cells
- Posoleucel and Placebo (Experimental): Arm 2: Regimen B
  Interventions: Biological: Posoleucel (formerly known as ALVR105) cells; Biological: Placebo (visually identical to Posoleucel)
- Placebo (Placebo Comparator): Arm 3: Regimen A
  Interventions: Biological: Placebo (visually identical to Posoleucel)

INTERVENTIONS:
Biological: Posoleucel (formerly known as ALVR105) cells — Infusion
  Arms: Posoleucel; Posoleucel and Placebo
Biological: Placebo (visually identical to Posoleucel) — Infusion
  Arms: Placebo; Posoleucel and Placebo

SUMMARY:
The purpose of this study is to compare Posoleucel (formerly known as ALVR105; Viralym-M) to placebo in kidney transplant recipients who have high or low levels of BK virus in their blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a kidney transplant performed greater than or equal to 28 days prior to enrollment
* At least 1 identified, suitably matched Posoleucel (ALVR105) cell line for infusion is available.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Undergone allogeneic hematopoietic cell transplantation
* Evidence or history of graft versus host disease (GVHD) or cytokine release syndrome (CRS).
* Uncontrolled or progressive bacterial or fungal infections
* Known or presumed pneumonia
* Ongoing therapy with high-dose systemic corticosteroids (ie, prednisone dose >0.5 mg/kg/day or equivalent).
* Pregnant or lactating or planning to become pregnant.
* Weight <40 kg.
* Patients who received, or planned to receive abatacept or belatacept, within 3 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Keck Medical Center of USC, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Piedmont Hospital, Atlanta, Georgia
  - Northwestern University Transplant Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - Tulane University School of Medicine, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - John Hopkins Hospital, Baltimore, Maryland
  - Harvard Medical School - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Erie County Medical Center, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Weil Medical College - NY Presbyterian Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - University of Cincinnati Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - UPMC Pinnacle-Harrisburg Hospital, Harrisburg, Pennsylvania
  - UPMC Montefiore Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Medical Center, Falls Church, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tzannou I, Papadopoulou A, Naik S, Leung K, Martinez CA, Ramos CA, Carrum G, Sasa G, Lulla P, Watanabe A, Kuvalekar M, Gee AP, Wu MF, Liu H, Grilley BJ, Krance RA, Gottschalk S, Brenner MK, Rooney CM, Heslop HE, Leen AM, Omer B. Off-the-Shelf Virus-Specific T Cells to Treat BK Virus, Human Herpesvirus 6, Cytomegalovirus, Epstein-Barr Virus, and Adenovirus Infections After Allogeneic Hematopoietic Stem-Cell Transplantation. J Clin Oncol. 2017 Nov 1;35(31):3547-3557. doi: 10.1200/JCO.2017.73.0655. Epub 2017 Aug 7. PMID 28783452
- [Background] Chandraker A, Regmi A, Gohh R, Sharma A, Woodle ES, Ansari MJ, Nair V, Chen LX, Alhamad T, Norman S, Cibrik D, Singh M, Alper A, Jain D, Zaky Z, Knechtle S, Sharfuddin A, Gupta G, Lonze BE, Young JH, Adey D, Faravardeh A, Dadhania DM, Rossi AP, Florescu D, Cardarelli F, Ma J, Gilmore S, Vasileiou S, Jindra PT, Wojciechowski D. Posoleucel in Kidney Transplant Recipients with BK Viremia: Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial. J Am Soc Nephrol. 2024 May 1;35(5):618-629. doi: 10.1681/ASN.0000000000000329. Epub 2024 Mar 12. PMID 38470444
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091
- [Derived] Vasileiou S, Kuvalekar M, Velazquez Y, Watanabe A, Leen AM, Gilmore SA. Phenotypic and functional characterization of posoleucel, a multivirus-specific T cell therapy for the treatment and prevention of viral infections in immunocompromised patients. Cytotherapy. 2024 Aug;26(8):869-877. doi: 10.1016/j.jcyt.2024.03.012. Epub 2024 Mar 19. PMID 38597860

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 26 sites in the United States between March 2021 and October 2022.
Pre-assignment Details: A total of 82 participants were screened during a 2-week screening period, of which 61 were randomized and received treatment.
Groups:
- Posoleucel (PSL) Group 1: Participants received PSL at a dose of 4 × 10^7 cells as a slow push intravenous (IV) infusion once per week for 3 weeks, then once every 14 days during the 12-week dosing period (8 total doses of PSL). Participants continued to be observed for a 12-week follow-up.
- PSL Group 2: Participants received PSL at a dose of 4 × 10^7 cells as a slow push IV infusion once per week for 3 weeks, then once every 28 days during the 12-week dosing period (5 total doses of PSL). Participants continued to be observed for a 12-week follow-up.
- Placebo: Participants received placebo matching PSL as a slow push IV infusion once per week for 3 weeks, then once every 14 days during the 12-week dosing period (8 total doses of placebo). Participants continued to be observed for a 12-week follow-up.
Period: Overall Study
Arm/Group | Posoleucel (PSL) Group 1 | PSL Group 2 | Placebo
Started | 20 | 22 | 19
Completed | 20 | 20 | 18
Not Completed | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: Included all randomized participants.
Groups:
- PSL Group 1: Participants received PSL at a dose of 4 × 10^7 cells as a slow push IV infusion once per week for 3 weeks, then once every 14 days during the 12-week dosing period (8 total doses of PSL). Participants continued to be observed for a 12-week follow-up.
- Total: Total of all reporting groups
Arm/Group | PSL Group 1 | PSL Group 2 | Placebo | Total
Number analyzed (Participants) | 20 | 22 | 19 | 61
Age, Continuous [Median (Full Range); unit: years] | 59.0 [21 to 75] | 54.0 [28 to 72] | 59.0 [47 to 75] | 58.0 [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 12
  Male | 17 | 17 | 15 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 2 | 9
  Not Hispanic or Latino | 18 | 17 | 17 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 3 | 5 | 9
  Black or African American | 4 | 9 | 4 | 17
  White | 12 | 7 | 10 | 29
  Other | 3 | 2 | 0 | 5
  Missing | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 19 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs are defined as AEs with a start date and time on or after the first dose of study treatment through the end of study.
  Clinically significant changes in vital signs, physical exams, laboratory assessments and electrocardiograms were also reported as TEAEs.
Time Frame: Day 1 to Week 24
Population: Safety Population: Included all participants who received any amount of PSL or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | PSL Group 1 | PSL Group 2 | Placebo
Number analyzed (Participants) | 20 | 22 | 19
Participants | 17 | 17 | 16

2. Secondary Outcome: Change From Baseline in BK Viral Load
Description: BK viral load was quantitated using polymerase chain reaction assays at the central laboratory. A negative change from baseline represents a reduction in BK viral load.
Time Frame: Baseline and Week 24
Population: ITT Population: Included all randomized participant with Week 24 BK viral load data available.
Measure: Median (Full Range); unit: log10 copies/mL
Arm/Group | PSL Group 1 | PSL Group 2 | Placebo
Number analyzed (Participants) | 19 | 19 | 17
log10 copies/mL | -0.830 [-2.08 to 0.11] | -0.520 [-3.55 to 0.52] | -0.330 [-2.08 to 0.27]

ADVERSE EVENTS:
Time Frame: Day 1 to Week 24
Description: Safety Population: Included all participants who received any amount of PSL or placebo.
Arm/Group | PSL Group 1 | PSL Group 2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/22 | 0/19
Other Adverse Events (participants affected / at risk) | 16/20 | 16/22 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PSL Group 1 (N=20) | PSL Group 2 (N=22) | Placebo (N=19)
Transplant rejection (Immune system disorders) | 0 | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Renal tuberculosis (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PSL Group 1 (N=20) | PSL Group 2 (N=22) | Placebo (N=19)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2
Pyrexia (General disorders) | 1 | 2 | 0
Chills (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 1
Pain (General disorders) | 1 | 0 | 1
Infusion site bruising (General disorders) | 0 | 1 | 0
Infusion site pain (General disorders) | 0 | 0 | 1
Injection site swelling (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Transplant rejection (Immune system disorders) | 2 | 0 | 0
COVID-19 (Infections and infestations) | 3 | 2 | 3
Epstein-Barr viraemia (Infections and infestations) | 2 | 0 | 1
Polyomavirus viraemia (Infections and infestations) | 2 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Polyomavirus-associated nephropathy (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
JC virus infection (Infections and infestations) | 0 | 1 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 1
Root canal infection (Infections and infestations) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1 | 0
Blood pressure diastolic decreased (Investigations) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0
Cystatin C increased (Investigations) | 0 | 1 | 0
Epstein-Barr virus test positive (Investigations) | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Heart rate decreased (Investigations) | 0 | 1 | 0
Immunosuppressant drug level increased (Investigations) | 0 | 1 | 0
JC polyomavirus test positive (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 4 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Post micturition dribble (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Urethral disorder (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hair disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/84/NCT04605484/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT04605484/SAP_001.pdf